CLINICAL TRIAL: NCT01159522
Title: A Phase 1 Dose Escalation Study of SCB01A in Subjects With Advanced Solid Tumors Who Have Failed Standard Therapy
Brief Title: A Dose Escalation Study of SCB01A in Subjects With Advanced Solid Tumors Who Have Failed Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SynCore Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCB01A-01
Record Dates: First submitted 2010-06-23; First posted 2010-07-09 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2015-09

CONDITIONS: Solid Tumors
Keywords: Advanced Solid Tumors Who Have Failed Standard Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCB01A (Experimental): This is an open-label, single-arm, dose-escalation, safety and tolerability study. Eligible subjects will be assigned to a SCB01A dose level at the time of study entry and scheduled to receive two treatment cycles with SCB01A for the observation of DLT. A treatment cycle is defined as a three-hour infusion of SCB01A given every 21 days. Unless any off-study criteria are met, the study period of each subject can be up to two cycles.
  Interventions: Drug: SCB01A

INTERVENTIONS:
Drug: SCB01A — This is an open-label, single-arm, dose-escalation, safety and tolerability study. Eligible subjects will be assigned to a SCB01A dose level at the time of study entry and scheduled to receive two treatment cycles with SCB01A for the observation of DLT. A treatment cycle is defined as a three-hour infusion of SCB01A given every 21 days. Unless any off-study criteria are met, the study period of each subject can be up to two cycles.

SUMMARY:
The goal of this study with SCB01A is to determine the Maximum Tolerated Dose of SCB01A in patients with advanced solid tumors that have failed previous therapy.

DETAILED DESCRIPTION:
This is an open-label, single-arm, dose-escalation, safety and tolerability study. Eligible subjects will be assigned to a SCB01A dose level at the time of study entry and scheduled to receive two treatment cycles with SCB01A for the observation of DLT. A treatment cycle is defined as a three-hour infusion of SCB01A given every 21 days. Unless any off-study criteria are met, the study period of each subject can be up to two cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are at least 18 years of age.
2. Have provided written informed consent prior to the initiation of study procedures.
3. Have histologically or cytologically confirmed diagnosis of an advanced solid tumor that has failed to respond to all available standard treatments.
4. Have ECOG PS scale of 0-1 at the time of enrollment.
5. Have adequate organ function:

   1. Bone marrow function:

      * White blood cell count (WBC) ≥ 4000/μL
      * Absolute neutrophil count (ANC) ≥ 1500/μL
      * Hemoglobin ≥ 10.0 g/dL
      * Platelet count ≥ 100,000/μL
   2. Hepatic Function:

      * Serum total bilirubin level ≤ 1.0 x upper normal limit
      * Serum alanine aminotransferase (ALT) level ≤ 2.5 x upper normal limit
   3. Renal Function:

      • Serum creatinine ≤ 1.0 x upper normal limit and creatinine clearance (estimated by Cockcroft-Gault formula) > 60 mL/min
   4. Heart Function:

      * Ejection fraction ≥ 55%
      * QTC < 450 msec
6. Have a life expectancy of at least 3 months
7. Have negative serum pregnancy test within 1 week before study drug administration (for women of childbearing potential and not diagnosed as germ cell tumor with beta-HCG only).
8. Are willing to practice medically accepted contraception (if the risk of contraception exists) throughout the study period (from screening until Final Visit).

Exclusion Criteria:

1. Subjects who have failed to recover from prior anti-cancer treatment-related toxicities, e.g. surgery, chemotherapy, radiotherapy, target therapy, biologic therapy, immunotherapy, alternative medicine, hormonal therapy, or investigational agent(s).
2. Treatment with an investigational drug, chemotherapy, targeting agent(s), biologic therapy (e.g., IL-2, Interferon, etc.), immunotherapy (e.g. tumor vaccine, etc.), alternative medicine or hormonal therapy (e.g. anti-estrogens, anti-androgens, etc.), radiation (except to bone) or surgery (except exploratory biopsy or intravenous device implantation, etc.) within 28 days prior to study entry.
3. Grade 2 or higher sensory neuropathy of any etiology.
4. Subjects with severe cardiopulmonary diseases (including history of stable, effort-induced or unstable angina pectoris, myocardial infarction, or arrhythmia) or other systemic diseases under poor control.
5. Females who are pregnant, lactating, or have a positive serum pregnancy test except those are diagnosed as germ cell tumor with beta-HCG prior to study treatment. Pre-menopausal women who are not abstinent must prove surgical sterility or compliance with a contraceptive regimen. Male subjects and male partners of female subjects must be abstinent, surgically sterile, or utilizing a barrier contraceptive method.
6. Tumor with central nervous system (CNS) involvement.
7. Subjects with concomitant active 2nd primary malignancies or disease-free for no more than 3 years following a definitive therapy for prior metachronous malignancies, except for surgically cured carcinoma, i.e. in situ of the cervix or adequately treated basal cell carcinoma of the skin or Dukes' A colorectal cancer.
8. Known history of allergy to any component of this investigational preparation.
9. History of exposure to SCB01A or its analogs.
10. Active infection requiring antibiotic therapy at time of study entry.
11. Is unwilling or unable to comply with the protocol requirements.
12. Known human immunodeficiency virus (HIV) infection.
13. History of receiving organ transplantation or immunologic illness that require continuous immunosuppressant agent therapy.
14. Have other medical or psychological conditions that would not permit the study participant to complete the study or sign informed consent.
15. Have any other disease, dysfunction, alcohol or drug abuse, physical examination or lab finding that, in the investigator's opinion, would exclude the subject from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD)in subjects with advanced solid tumor | Each subject can be given up to 2 cycles of SCB01A. Each cycle will be 21 days.
  MTD is the dose at which at least two subjects experience the DLT; and DLT is defined as Grade 3 or greater Neutropenia, Thrombocytopenia, prolonged QTc, non-hematological adverse events and neurotoxicity
To determine DLT (Dose Limiting Toxicity) in subjects with advanced solid tumor | Each subject can be given up to 2 cycles of SCB01A. Each cycle will be 21 days.
  DLT is defined as Grade 3 or greater Neutropenia, Thrombocytopenia, prolonged QTc, non-hematological adverse events and neurotoxicity

SECONDARY OUTCOMES:
Safety will be evaluated by physical examinations, vital signs, laboratory assessments, ECOG PS scale, and the incidence and severity of adverse events. | ECOG-PS, AE's, physical examinations, vital signs, laboratory assessments will be assessed weekly.
For PK profile, blood samples will be collected at various time points | PK blood samples will be taken immediately pre-infusion then at 1, 2, 3, 4, 6, 10, 21 and 24 hours after start of infusion on Day 1
Tumor response will be assessed by RECIST v1.1 | During screening and final visit

CONTACTS AND LOCATIONS:
Overall Officials: Muh-Hwan Su, Ph.D., Study Director — SynCore Biotechnology
Locations (3):
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei

REFERENCES:
- [Derived] Shiah HS, Chiang NJ, Lin CC, Yen CJ, Tsai HJ, Wu SY, Su WC, Chang KY, Wang CC, Chang JY, Chen LT. Phase I Dose-Escalation Study of SCB01A, a Microtubule Inhibitor with Vascular Disrupting Activity, in Patients with Advanced Solid Tumors. Oncologist. 2021 Apr;26(4):e567-e579. doi: 10.1002/onco.13612. Epub 2020 Dec 18. PMID 33245172